CLINICAL TRIAL: NCT06627582
Title: Persistent Postmastectomy Pain: Defining the Burden of Disease and the Role of Surgical Reinnervation in Patients With Breast Reconstruction
Brief Title: A Study on Pain After Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-271
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Mastectomy; Mastectomy Patient; Mastectomy and Breast Reconstruction; Breast Reconstruction; Breast Reconstruction After Mastectomy; Postmastectomy Pain
Keywords: Postmastectomy Pain; breast reconstruction after mastectomy; breast reconstruction; mastectomy and breast reconstruction; mastectomy; mastectomy patient; 24-271; Memorial Sloan Kettering Cancer Center

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postmastectomy Reconstruction Participants (Experimental): Participants will be postmastectomy reconstruction and >/= 6 months postoperative
  Interventions: Behavioral: PROMIS Scale v2.0 - Pain Intensity 3a; Behavioral: PROMIS 29+2; Behavioral: PROMIS Scale v2.0 - Nociceptive Pain Quality 5a; Behavioral: PROMIS Scale v2.0 - Neuropathic Pain Quality 5a

INTERVENTIONS:
Behavioral: PROMIS Scale v2.0 - Pain Intensity 3a — PROMIS Scale v2.0 - Pain Intensity 3a is a 3-question short form in which patients rate their worst, average, and current level of pain during the past 7 days.
Behavioral: PROMIS 29+2 — PROMIS 29+2 (PROMIS-Preference, PROPr) is a compilation of item banks to assess pain intensity
Behavioral: PROMIS Scale v2.0 - Nociceptive Pain Quality 5a — 5-question short form that identifies patients who have experienced nociceptive pain during the past 7 days
Behavioral: PROMIS Scale v2.0 - Neuropathic Pain Quality 5a — 5-question short form that identifies patients who have experienced neuropathic pain during the past 7 days

SUMMARY:
The purpose of this study is to find out how common persistent postmastectomy pain (PPMP) is among people who have had a mastectomy and breast reconstruction surgery for their breast cancer. The study will also look at how effective regenerative peripheral nerve interface (RPNI) surgery is for reducing pain from neuropathic PPMP after breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥18 years
* History of mastectomy for breast cancer or genetic predisposition to breast cancer
* History of breast reconstruction with implants and/or autologous tissue
* At least 6 months of follow-up after reconstruction
* Patient treated at MSK

Exclusion Criteria:

* Exchange or revision surgery within 6 months
* Active medical reason for pain (e.g., infectious, neoplastic, wound related)
* Greater than 15 years post-reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Persistent Postmastectomy Pain | up to 6 months
  The primary objective is to estimate the prevalence of Persistent Postmastectomy Pain/PPMP in breast cancer survivors treated with mastectomy and reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Rochlin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org